CLINICAL TRIAL: NCT05979870
Title: Artificial Intelligence in New Cardiac MR Markers for Congenital Heart Disease -Improving the Assessment, Monitoring and Prediction in Children
Brief Title: Artificial Intelligence in New Cardiac MR Markers for Congenital Heart Disease
Acronym: AI-CMR
Status: Enrolling by invitation | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Charlotte de Lange, MD Associate Professor, senior consultant, Sahlgrenska University Hospital
Other Study IDs: 277238
Record Dates: First submitted 2023-07-31; First posted 2023-08-07 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Aortic Valve Disease; Pulmonary Valve Disease; Child, Only; Magnetic Resonance Imaging; Risk Stratification
MeSH Terms: conditions — Aortic Valve Disease | interventions — Balloon Valvuloplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood, serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Aortic valve disease-operation: Surgery of the aortic valve:
  Cardiac and blood flow changes assessed by advanced MRI methods before and after treatment.
  Interventions: Procedure: Valvuloplasty,
- Aortic valve disease-intervention: Interventional treatment of the aortic valve:
  Cardiac and blood flow changes assessed by advanced MRI methods before and after treatment.
  Interventions: Procedure: Valvuloplasty,
- Pulmonary valve disease-operation: Surgery of the pulmonary valve:
  Cardiac and blood flow changes assessed by advanced MRI methods before and after treatment.
  Interventions: Procedure: Valvuloplasty,
- Pulmonary valve disease-intervention: Interventional treatment of the pulmonary valve:
  Cardiac and blood flow changes assessed by advanced MRI methods before and after treatment
  Interventions: Procedure: Valvuloplasty,

INTERVENTIONS:
Procedure: Valvuloplasty, — Choice of type of intervention decided on a multidisciplinary conference
  Other Names: surgical valvular repair

SUMMARY:
The goal of this study is to investigate children with aortic and pulmonary valve disease treated or untreated longitudinally. Established CMR measures with additional newly developped, promising, highly refined and clinically applicable quantitative imaging biomarkers, will be utilized as compared to the conventional CMR estimates.

The main question[s] it aims to answer are:

* [question 1]To evaluate risk stratification for surgery and intervention of the aortic- and pulmonary valve
* [question 2]Investigate the cardiac and vascular hemodynamic and morphological changes before and after interventional or surgical treatment of the aortic- and pulmonary valve at short and long term.

Participants will undergo cardiac MRI before and after interventional or surgical treatment of the aortic or pulmonary valve Researchers will compare MRI data to an age matched control group established at the department in another study.

DETAILED DESCRIPTION:
Background:

An increasing number of children with complex congenital heart disease (CHD) are today treated and survive into adulthood. They are in need of a lifelong surveillance for cardiovascular complications and an individualised treatment.

In paediatric aortic and pulmonary valve disease, the long-term complications are related to valvular dysfunction with myocardial fibrosis and ventricular dysfunction as a result of longstanding volume or pressure overload. Many patients will need surgery or interventional treatment already in childhood, where the optimal timing of the intervention is crucial, since early treatment may prevent irreversible injury to the heart.

Moreover, to enable detection of recurrent or new problems early, a long-term diagnostic follow-up is needed where cardiovascular magnetic resonance (CMR) has become important for a serial reproducible assessment of morphology, function and recently advanced methods for flow and tissue characterisation. Still the the clinical decision of the perfect time-point and type of treatment for a child, may be difficult in many cases, and better measures are needed.

Aim:

This project will investigate children with aortic and pulmonary valve disease treated or untreated longitudinally using established CMR measures with additional newly developed, promising, highly refined and clinically applicable quantitative imaging biomarkers, as compared to the conventional CMR estimates. Investigators aim to evaluate risk stratification and investigate the haemodynamic and morphological changes as well as physical capacity before and after interventional or surgical treatment at short and long term.

CMR will be analysed for established imaging biomarkers as well as the potential value of new data-driven computer tools searching for new information in the CMR images i.e. shape/texture analysis of tissue change, regional haemodynamics, blood flow in relation to metallic implants and evaluation of myocardial deformation over time.

CMR measures will be compared to data from echocardiography, catheterization and serological markers.

Clinical importance:

If the new refined CMR biomarkers can reveal improved disease characterisation, they may reveal feasible in aiding the clinical decision making to optimise timing of intervention and predicting long term complications. This could contribute to individualise the treatment and improve health in children with CHD. The study may lead to improved patient care and use of socio-economical resources.

ELIGIBILITY:
Inclusion Criteria:

* aortic valve disease
* or pulmonary valve disease
* clinical indication for valvular surgery
* or clinical indication for valvular intervention

Exclusion Criteria:

* contraindications for MRI
* need of sedation or general anesthesia, unless there is a clinical indication for a CMR

Ages: 1 Week to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Childen aged 0-18 years old with aortic or pulmonary valve disease in need of treatment admitted to the Paediatric Heart Centre, Queen Silvia Childrens' Hospital, Gothenburg Sweden.
  Patients will be invited to participate in the study after a multidisciplinary conference on decision of treatment
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
CMR measures | Before and after 6 months, 1 year and up to 3 years after intervention or surgery
  Measurement by CMR of changes in ventricular function, remodelling, tissue characterisation and advanced four dimensional flow (4D-flow) measurements after surgery or intervention
Physical capacity | Before and after 6 months, 1 year and up to 3 years after intervention or surgery
  Measurement of physical capacity after surgery or intervention, by cardiopulmonary exercise testing (CPET)

SECONDARY OUTCOMES:
CMR derived flow measurements near metallic implants, stents | after 6 months, 1 year and up to 3 years after intervention
  Refined measurements of CMR derived 4D-flow measurements near metallic implants, stents

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte de Lange, MD, Assoc. Prof, Principal Investigator — Sahlgrenska University hospital, Queen Silvia Childrens' Hospital
Locations (1):
- Queen Silvia Children'sHospital, Sahlgrenska University Hospital, Gothenburg, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided